CLINICAL TRIAL: NCT00991900
Title: Short Term and Day to Day Reproducibility of Reflectometric Measurement of Retinal Oxygen Saturation in Healthy Subjects
Status: Withdrawn | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Ass.Prof.Dr.med., Medical University of Vienna
Other Study IDs: OPHT-030409
Record Dates: First submitted 2009-10-07; First posted 2009-10-08 (Estimated); Last update posted 2018-06-11 (Actual); Status verified 2018-06

CONDITIONS: Ocular Physiology

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Healthy subjects
  Interventions: Device: Measurement of oxygen saturation of retinal vessels with optical reflectometer

INTERVENTIONS:
Device: Measurement of oxygen saturation of retinal vessels with optical reflectometer — 5 repeated measurements on both study days

SUMMARY:
Adequate perfusion and oxygenation is essential for the function of the inner retina. Although this is a well known fact, measurement of oxygen saturation in the eye is still a delicate and not fully explored task. However, recently a new instrument for the non-invasive measurement of retinal vessel oxygen saturation has been introduced. Unfortunately, no data about reproducibility in humans is yet available for this instrument. Consequently, the current study seeks to evaluate the short term and day to day reproducibility of retinal vessel oxygenation in healthy volunteers.

20 healthy volunteers will be included and oxygen saturation of retinal vessels will be determined. The reproducibility of the results will be tested by repeated measurements and the collected data will be independently analyzed by two observers.

ELIGIBILITY:
Inclusion Criteria:

* Men and Women aged between 18 and 35 years,
* Nonsmokers
* Body mass index between 15th and 85th percentile
* Normal ophthalmic findings, ametropia < 3 Dpt.

Exclusion Criteria:

* Regular use of medication, abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study
* Treatment in the previous 3 weeks with any drug except oral contraceptives
* Symptoms of a clinically relevant illness in the 3 weeks before the study day
* Blood donation during the previous 3 weeks

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 20 healthy volunteers will be included.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-08; Primary Completion 2009-10 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Coefficients of variation of oxygen measurement | 5 measurements on both study days

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria